CLINICAL TRIAL: NCT02864485
Title: Assessment of a Protocol Using a Combination of Neo-adjuvant Chemotherapy Plus Living Donor Liver Transplantation for Non-Resectable Liver Metastases From Colorectal Cancer
Brief Title: Living Donor Liver Transplantation for Unresectable Colorectal Cancer Liver Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-9382-C
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Live donor liver transplantation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- transplantation (Experimental): Live donor liver transplantation for the treatment of unresectable colorectal cancer liver metastases
  Interventions: Procedure: live donor liver transplantation

INTERVENTIONS:
Procedure: live donor liver transplantation — live donor liver transplantation

SUMMARY:
Patients with unresectable liver metastases (LM) from colorectal cancer (CRC)have a poor prognosis. In patients with resectable disease, surgery offers a distinct survival benefit. This study will offer live donor liver transplantation (LDLT) to select patients with unresectable metastases that are 1) limited to the liver and 2) stable (non-progressing) on standard chemotherapy. Potential participants will be evaluated for liver transplant suitability and must also have a willing, healthy living donor come forward for evaluation. Those participants who undergo LDLT will be followed for survival, disease-free survival and quality of life for 5 years and compared to a "control group" of participants who drop out of study prior to transplantation due to reasons other than cancer progression.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a leading cause of cancer-related mortality worldwide. Approximately half of all patients develop metastases, often to the liver or lung. Surgical treatment of liver metastases (LM) is the only curative treatment option; however, it has been estimated that only 20-40% of patients are candidates for liver resection. Surgery offers a distinct survival advantage: the 5-year survival after liver resection for LM is around 40-50% in most studies versus 10-20% 5-year survival for chemotherapy alone.

In cases where the colorectal metastases are isolated to the liver but "unresectable", the total hepatectomy resulting from liver transplantation would remove all evident disease. CRC LM are considered an absolute contraindication for liver transplantation (LT) at most centers but recent reports of LT for colorectal LM from a single center in Oslo, Norway demonstrated a 5-year survival of 56%. The Norway study was not stringent about inclusion criteria or pre-transplant chemotherapy, and transplanted patients whose tumors were actively growing. As a result many participants developed disease recurrence quite rapidly following transplant. The investigators hypothesize that tighter criteria would result in improved outcomes.

Unfortunately, with a lack of deceased donor grafts for the investigators existing transplant patients, the investigators cannot utilize decease donor grafts for this study. Therefore the investigators will explore Living Donor Liver Transplantation (LDLT). Furthermore, LDLT is an elective surgery, allowing for more control over pre-transplant chemotherapy and tumor monitoring. This study will offer live donor liver transplantation (LDLT) to select patients with unresectable metastases that are 1) limited to the liver and 2) stable (non-progressing) on standard chemotherapy. Potential participants will be evaluated for liver transplant suitability and must also have a willing, healthy living donor come forward for evaluation. Those participants who undergo LDLT will be followed for survival, disease-free survival and quality of life for 5 years and compared to a "control group" of participants who drop out of study prior to transplantation due to reasons other than cancer progression.

ELIGIBILITY:
Inclusion Criteria:

* Must reside in Canada
* ECOG ( Eastern Cooperative Oncology Group) score : 0-1 at all times prior to LDLT (excursions to ECOG 2 allowed at investigator's discretion)
* Proven colorectal Liver Metastases (LM).
* Willing and able to provide written informed consent.
* Negative serum pregnancy test for women of childbearing potential
* Both men and women must agree to use adequate barrier birth control measures during the course of the trial.
* At least 1 "acceptable", ABO-compatible living donor has stepped forward
* Primary Colorectal cancer tumor stage is ≤T4a
* Time from primary CRC resection to transplant is ≥6 months
* Bilateral and non-resectable LM
* No major vascular invasion by LM; metastases isolated to liver
* The patient has undergone systemic chemotherapy (eg. FOLFOX +/- bevacizumab or FOLFIRI +/- bevacizumab) for ≥3 months
* demonstrated stability or regression of LM over at minimum the 3 months preceding screening
* Carcinoembryonic Antigen (CEA) values are stable or decreasing at all timepoints prior to the transplant surgery.

Exclusion Criteria:

* Previous or concurrent cancer (with some exceptions)
* prior lung resection
* Progression of LM at any timepoint prior to transplant surgery
* Renal dysfunction with an estimated creatinine clearance of less than 50 ml/min
* Pulmonary insufficiency
* History of cardiac disease
* Known history of human immunodeficiency virus (HIV) infection or chronic hepatitis B and/or C infection.
* Patients with debilitating neuropathy. (CTCAE > grade 2)
* BRAF + tumors
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
patient survival | 5 years
disease-free survival | 5 years

SECONDARY OUTCOMES:
patterns of cancer recurrence after liver transplantation | 5 years
types of cancer recurrence treatments | 5 years
Number of participants that drop out of study prior to receiving intervention (transplantation surgery) due to chemotherapy-related adverse events, as assessed by CTCAE v4.0 | prior to liver transplantation
self-reported quality of life as assessed by EORTC QLQ-C30 questionnaire | 6 month intervals for 5 years
  Compare the QoL of participants undergoing intervention vs participants that drop-out (for non cancer related reasons and are thereafter receiving palliative chemotherapy)
survival of intervention vs standard treatment | 1-, 3- and 5 years
  Compare the 1-, 3- and 5- year survival of patients that undergo intervention with those that drop-out of the study (due to non-cancer related reasons and receive standard chemotherapy)
patient survival | 1 year
patient survival | 3 years
disease-free survival | 1 year
disease-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Sapisochin, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Rajendran L, Claasen MP, McGilvray ID, Cattral MS, Ghanekar A, Selzner N, Burkes R, Winter E, Gallinger S, Sapisochin G. Toronto Management of Initially Unresectable Liver Metastasis from Colorectal Cancer in a Living Donor Liver Transplant Program. J Am Coll Surg. 2023 Aug 1;237(2):231-242. doi: 10.1097/XCS.0000000000000734. Epub 2023 May 3. PMID 37130158